CLINICAL TRIAL: NCT06271304
Title: Stabilizing Mood and Sleep With Blue Blocking Eyewear in Bipolar Disorder
Acronym: BLUES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLUES
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Outcome assessors will be blinded to the treatment assignment. At the beginning of each assessment, participants will be instructed not to describe or discuss their glasses with the assessor. Because the two types of glasses are of different color (clear (LF) and orange (BB)), we cannot guarantee a full blinding of the participants. Participants will be informed that we are studying the effects of two different types of light filters without more detail so they will not be provided with certain knowledge of which condition is expected to yield the largest effect. We will assess the integrity of the blind by asking participants whether they think they received glasses with high or low filtration lenses at the end of the study. Participants will be discouraged from actively seeking information about sleep glasses during the study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are instructed not to discuss the appearance of their designated eyewear with their care providers or the investigator or outcome assessor. Participants are not informed of the exact filtration level of their eyewear.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue blocking glasses (BB) (Experimental): Eyewear with orange-tinted lenses that block 99% of short wavelength visible light < 500 nm
  Interventions: Device: Blue blocking eyewear
- Low filtration glasses (LF) (Sham Comparator): Eyewear with clear lenses that block 15% of short wavelength light < 500 nm
  Interventions: Device: Low filtration eyewear

INTERVENTIONS:
Device: Blue blocking eyewear — Eyewear is worn daily from 6 PM to 8 AM during manic/hypomanic state Eyewear is worn daily 2 hours before planned bedtime during euthymic, depressive and mixed state
  Arms: Blue blocking glasses (BB)
Device: Low filtration eyewear — Eyewear is worn daily from 6 PM to 8 AM during manic/hypomanic state Eyewear is worn daily 2 hours before planned bedtime during euthymic, depressive and mixed state
  Arms: Low filtration glasses (LF)

SUMMARY:
The study investigates whether add-on treatment with eyewear that blocks the short wavelengths of visible light (<500nm) reduces manic symptoms and improves sleep in patients receiving outpatient treatment as usual for bipolar disorder.

When in a hypomanic or manic phase, participants will be randomized to receive add-on treatment with either blue blocking or low filtration eyewear from 18 PM to 8 AM daily for 7 days.

After this initial intervention phase, the eyewear is used daily for 3 months in either antimanic dose (14 hours) or maintenance dose (2 hours before bedtime).

DETAILED DESCRIPTION:
The study is a 2-arm single-blind RCT to assess the effects of blue blocking (BB) or clear glasses as an acute 7-day antimanic intervention and as a 3-month mood stabilizing maintenance intervention. BB or clear glasses will be applied in addition to outpatient TAU for BD. Participants will be recruited among patients treated for BD in specialized outpatient clinics within the Mental Health Center Copenhagen.

The active intervention is BB-glasses that eliminate 99 % of light with a wavelength below 530 nm, whereas the clear glasses filter out only 15% of short wavelength light (low filtration (LF).

Participation includes 3 months use of the designated eyewear along with daily electronic self-monitoring of mood, sleep and activity as well as participation in a 2-day baseline assessment and a total of 3 follow-up visits including clinical assessment interview, questionnaires, and actigraphic (48 hours) and pupillometric assessments at day 9, week 5 and week 15.

Participants will be included during hypomanic or manic state and begin treatment with an antimanic dosage of 14 hours (6 PM - 8 AM) for 7 consecutive days. Subsequently, during the 3-month follow-up period, the dosage (hours using the glasses) can be adjusted according to the current state, with use for 14 hours during hypomanic/manic phases and 2 hours before bedtime during euthymic and depressive states.

Outcome assessors will be blinded to the treatment assignment and patients will be informed that they are randomized to eyewear with either high or low filtration of light. Patients will be randomized on a 1:1 basis with stratification according to sex and outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder
* YMRS-score >13
* Age 18-60 years
* Speaks and writes Danish at a level equal to mother tongue

Exclusion Criteria:

* Not willing or able to adhere to the protocol
* Severe eye disorder or eye trauma
* Treatment with betablockers
* Sleep disturbances not related to BD (e.g, sleep apnea, restless legs syndrome) • • Substance abuse
* Unwilling to use the electronic self-monitoring system, the Monsenso system
* Prior/current use of BB glasses
* Current/planned pregnancy
* Night shift work
* Suicidality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Manic symptoms | 7 days
  Change in Young Mania Rating Scale Score, range 0-60, higher scores indicating greater manic symptom load

SECONDARY OUTCOMES:
Mood instability | 15 weeks
  Change in day-to-day variation in electronically self-monitored mood scores
Objective sleep quality | 7 days
  Actigraphic measures of sleep latency, sleep time, efficiency and wake periods
Objective sleep quality | 15 weeks
  Actigraphic measures of sleep latency, sleep time, efficiency and wake periods
Subjective sleep quality | 7 days
  change in sleep scores from a modified version of the Pittsburgh Sleep Quality Index, range 0-21, higher scores indicating worse sleep quality
Subjective sleep quality | 15 weeks
  change in sleep scores from a modified version of the Pittsburgh Sleep Quality Index, range 0-21, higher scores indicating worse sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Lars Kessing, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No